CLINICAL TRIAL: NCT06623812
Title: Satiety Responses of Meals Consisting of Different Protein Sources
Brief Title: Alternative ProtEin Satiety Study (APES Study)
Acronym: APES
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Singapore Institute of Food and Biotechnology Innovation (Other Government)
Responsible Party: Principal Investigator, Teo Pey Sze, Senior Scientist I, Singapore Institute of Food and Biotechnology Innovation
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 2024-089
Record Dates: First submitted 2024-09-25; First posted 2024-10-02 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: Healthy Male Adults Participants
Keywords: Satiety; Alternative Protein; Protein Quality

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Animal Protein (Active Comparator): A standardized typical lunch test meal consists of an animal-based protein source (Animal Protein). The total weight of meal, total energy served, as well as energy from macronutrients are standardized across the three test meals.
  Interventions: Other: Behavioral: Post- meal satiety and subsequent ad-libitum meal energy intake
- Plant Protein 1 with lower DIAAS Score (lower protein quality) (Active Comparator): A standardized typical lunch test meal consists of a plant-based protein source with a lower DIAAS Score (Plant protein 1- lower protein quality). The total weight of meal, total energy served, as well as energy from macronutrients are standardized across the three test meals.
  Interventions: Other: Behavioral: Post- meal satiety and subsequent ad-libitum meal energy intake
- Plant Protein 2 with higher DIAAS Score (higher protein quality) (Active Comparator): A standardized typical lunch test meal consists of a plant-based protein source with a higher DIAAS Score (Plant protein 2- higher protein quality). The total weight of meal, total energy served, as well as energy from macronutrients are standardized across the three test meals.
  Interventions: Other: Behavioral: Post- meal satiety and subsequent ad-libitum meal energy intake

INTERVENTIONS:
Other: Behavioral: Post- meal satiety and subsequent ad-libitum meal energy intake — Investigate differences in post meal satiety and subsequent post meal energy intake after consuming fixed portion meals with different protein source and/ or different protein quality

SUMMARY:
This project aims to study the effects of different protein quality (i.e. high vs. low) and protein sources (i.e. plant protein vs. conventional animal protein) on post-meal satiety and satisfaction. The protein quality score of meals will be calculated using the published digestible indispensable amino acid score (DIAAS). The proposed study will investigate the link between protein quality, protein source, and the post-meal satiety responses, using a realistic lunch meal approach, in humans. Other than the self-reported visual analogue scale (VAS) satiety response, the postprandial glucose dips (i.e. 2-3hours post-meal) will be collected by continuous glucose monitoring (CGMS) as an objective indicator of postprandial self-reported hunger and subsequent energy intake. In addition, the oral processing behaviours of participants will be captured and compared between the test meals.

DETAILED DESCRIPTION:
Aim: To investigate how differences in protein quality (i.e. high vs low quality) and protein sources (i.e. plant vs animal proteins) influence the satisfaction, satiety responses (fullness over the time) and subsequent food intake.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male
* Aged between 21 and 50-year-old
* Are of normal weight (BMI 18-25kg/m2)
* Stable weight for the previous 12 months (<5kg weight fluctuation in the previous year)
* Healthy dentition and ability to bite, chew and swallow normally
* No history of pain or discomfort in jaw movements or excessive teeth clenching or grinding
* No dental carries or periodontal disease
* Own a mobile device with Apple iOS Operating System version 15.0 -17.3 or Android Operating System version 10-14
* Have access to a data plan
* Comfortable with needles and insertion of a Continuous Glucose Monitoring System device for 3-7 days

Exclusion Criteria:

* Are a smoker
* Have any dislikes, intolerances or allergies to foods or common food ingredients e.g. nuts, soya, wheat, gluten, cereal, fruits, biscuits, dairy products, rice, vegetable, meat, seafood, sugar and sweetener, gelatin, natural food colourings or flavourings (e.g. MSG), etc.
* Have any specific dietary requirements and/ or restrictions (e.g. Vegan/ vegetarian, religious beliefs, lactose intolerance, calorie restricted diet etc.)
* Known sensitivity to medical-grade adhesives
* Bleeding disorders (e.g Hemophilia, von Willebrand disease etc.)
* Have sinus problems that affect your taste and smell
* Have known glucose-6-phosphate dehydrogenase (G6PD) deficiency
* Are taking insulin or medication known to affect your appetite or metabolism
* Have major chronic diseases such as heart disease, cancer or diabetes mellitus etc.
* Have active Tuberculosis (TB) or currently receiving treatment for TB
* Have any known Chronic Infection or known to suffer from or have previously suffered from or is a carrier of Hepatitis B Virus (HBV), Hepatitis C Virus (HCV), Human Immunodeficiency Virus (HIV)
* Are a member of the research team or their immediate family members. Immediate family member is defined as a spouse, parent, child, or sibling, whether biological or legally adopted
* Are enrolled in a concurrent research study judged not to be scientifically or medically compatible with this study

Ages: 21 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Post-Prandial Sensor Glucose Readings | During the test day 2, 5, 8, up to 48 hours per test day. There is a one-week wash-out period between test days
  A continuous monitoring glucose sensor will be used to measure participants sensor glucose readings. The post-prandial sensor glucose readings 2-3h post meal will be used as an objective indicator of postprandial self-reported hunger and subsequent energy intake.
Oral processing behaviour | During test day 2, 5 and 8, up to 20 minutes per test day. There is a one-week wash-out period between test days
  Participants will be video recorded during the lunch sessions to measure oral processing behavior (e.g., derived from number of bites, chews, swallows and eating duration) of the fixed portion test meals using an annotation software
Change in Post breakfast satiety responses | During test day 2, 5 and 8, at 15- or 30-minutes intervals, up to 4 hours each test day. There is a one-week wash-out period between test days
  Participants will be asked rate their appetite sensations using a visual analogue scale (VAS) pre- and post meals. VAS is anchored at: Not at all (0) to Extremely (100), where a higher score will indicate greater intensity.
Ad-libitum snack intake | During test day 2, 5, and 8, up to 15 minutes per test day. There is a one-week wash-out period between test days
  Participants will be asked to eat an ad-libitum amount of snack 2h post lunch. The amount of food consumed will be weighed.
Subsequent food intake post test meal | During test day 2, 5 and 8, up to participant's bedtime per test day (before 12am midnight of the next day). There is a one-week wash-out period between test days
  Participants will be asked to bring a food dairy home to record their food and beverage intake for the rest of the test day. This is to assess participants calorie intake for the remaining day on the test session.
Change in Post lunch satiety responses | During test day 2, 5 and 8, at 15- or 30-minutes intervals, up to 2 hours each test day. There is a one-week wash-out period between test days
  Participants will be asked rate their appetite sensations using a visual analogue scale (VAS) pre- and post meals. VAS is anchored at: Not at all (0) to Extremely(100), where a higher score will indicate greater intensity.

CONTACTS AND LOCATIONS:
Overall Officials: Pey Sze Teo, PhD, Principal Investigator — Singapore Institute of Food and Biotechnology Innovation (SIFBI)

IPD SHARING:
Plan to Share IPD: No